CLINICAL TRIAL: NCT01150357
Title: A Multicenter, Randomized, Double-blind, 8 Week Study to Evaluate the Dose Response, Efficacy and Safety of Aliskiren in Pediatric Hypertensive Patients 6-17 Years of Age
Brief Title: Safety and Efficacy of Aliskiren in Pediatric Hypertensive Patients 6-17 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2365; 2009-017028-22 (EudraCT Number)
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension
Keywords: Pediatric hypertension; primary hypertension; secondary hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Low Dose Aliskiren (Experimental): Participants received body-weight stratified dose of aliskiren capsules (6.25/12.5/25 mg) once daily. Participants whose body weight ≥ 20 kilogram (kg) to less than < 50 kg received 6.25 mg; ≥50 kg and < 80 kg received 12.5 mg and ≥ 80 kg and ≤ 150 kg received 25 mg of aliskiren.
  Interventions: Drug: Aliskiren (6.25/12.5/25 mg)
- Mid dose (Experimental): Participants received body-weight stratified dose of aliskiren capsules (37.5/75/150 mg) once daily. Participants whose body weight ≥ 20 kg to < 50 kg received 37.5 mg; ≥50 kg and < 80 kg received 75 mg and ≥ 80 kg and ≤ 150 kg received 150 mg of aliskiren.
  Interventions: Drug: Aliskiren (37.5/75/150 mg)
- High dose (Experimental): Participants received body-weight stratified dose of aliskiren capsules (150/300/600 mg) once daily. Participants whose body weight ≥ 20 kg to < 50 kg received 150 mg; ≥50 kg and < 80 kg received 300 mg and ≥ 80 kg and ≤ 150 kg received 600 mg of aliskiren.
  Interventions: Drug: Aliskiren (150/300/600 mg)

INTERVENTIONS:
Drug: Aliskiren (6.25/12.5/25 mg) — Aliskiren dispensing capsules containing minitablets (3.125 mg per minitablet). For the low dose arm, participants used one or more of the 6.25 mg capsule (containing 2 minitablets) once daily to reach the body-weight stratified dose of aliskiren.
  Arms: Low Dose Aliskiren
Drug: Aliskiren (37.5/75/150 mg) — Aliskiren dispensing capsules containing minitablets (3.125 mg per minitablet). For the medium dose arm, participants used one or more of the 37.5 mg capsule (containing 12 minitablets) once daily to reach the body- weight stratified dose of aliskiren.
  Arms: Mid dose
Drug: Aliskiren (150/300/600 mg) — Aliskiren dispensing capsules containing minitablets (3.125 mg per minitablet). For the high dose arm, participants used one or more of the 150 mg capsule (containing 48 minitablets) once daily to reach the body- weight stratified dose of aliskiren.
  Arms: High dose

SUMMARY:
This double-blind 8 week study will evaluate dose response, efficacy (blood pressure lowering effect) and safety of aliskiren in children 6 - 17 years old with hypertension at low, mid and high weight-based doses. The low dose ranges from 6.25 mg to 25 mg of aliskiren, the mid dose ranges from 37.5 mg to 150 mg of aliskiren and the high dose ranges from 150 mg to 600 mg of aliskiren. This study is being conducted to support monotherapy registration of aliskiren for the treatment of hypertension in children 6-17 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of hypertension as defined in the NHLBI 4th Report, 2004
* msSBP (mean of 3 measurements) must be ≥ 95th percentile for age, gender and height, at Visit 2 (randomization) measurement as defined by the NHLBI 4th Report, 2004

Exclusion Criteria:

* Patient receiving immunosuppressant medication (e.g. cyclosporine, MMF, etc) other than oral/topical steroids, for any medical condition
* Current diagnosis of heart failure (NYHA Class II-IV) or history of cardiomyopathy or obstructive valvular disease
* msSBP ≥ 25% above the 95th percentile
* Second or third degree heart block without a pacemaker
* AST/SGOT or ALT/SGPT >3 times the upper limit of the reference range
* Total bilirubin > 2 times the upper limit of the reference range
* Creatinine clearance < 30 mL/min/1.73m² (calculated using Modified Schwartz formula to estimate glomerular filtration rate [GFR]), based on the serum creatinine concentration obtained at the screening visit)
* WBC count < 3000/mm³

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 267 (Actual)
Dates: Start 2010-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- United States (22):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Dalton, Georgia
  - Novartis Investigative Site, Lewiston, Idaho
  - Novartis Investigative Site, Park Ridge, Illinois
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Hattiesburg, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Hackensack, New Jersey
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Charleston, West Virginia
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Marburg, Germany
- Novartis Investigative Site, Guatemala City, Departamento de Guatemala, Guatemala
- Hungary (6):
  - Novartis Investigative Site, Nyíregyháza, Hungary
  - Novartis Investigative Site, Szeged, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Veszprém
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, San Juan, Puerto Rico
- Slovakia (5):
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Martin, Slovakia
  - Novartis Investigative Site, Myjava, Slovakia
  - Novartis Investigative Site, Prešov, Slovakia
  - Novartis Investigative Site, Trnava, Slovakia
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara, Turkey
  - Novartis Investigative Site, Izmir

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 51 centers in 8 countries.
Pre-assignment Details: A total of 334 participants were screened and placed in screening phase of single blind placebo washout period for up to a maximum of three weeks. Out of 334, 268 participants were randomized in Phase 1 including 1 mis-randomized participants who did not receive any medication. Therefore total of 267 was enrolled in this study
Groups:
- Aliskiren Low (6.25/12.5/25 mg): During Phase 1: Participants received body-weight stratified dose of aliskiren capsules (6.25/12.5/25 mg) once daily. Participants whose body weight ≥ 20 kilogram (kg) to less than < 50 kg received 6.25 mg; ≥50 kg and < 80 kg received 12.5 mg and ≥ 80 kg and ≤ 150 kg received 25 mg of aliskiren.
  During Phase 2: 50 participants continued the aliskiren treatment from Phase 1, while 57 participants switched to placebo treatment.
- Aliskiren Mid (37.5/75/150 mg): During Phase 1: Participants received body-weight stratified dose of aliskiren capsules (37.5/75/150 mg) once daily. Participants whose body weight ≥ 20 kg to < 50 kg received 37.5 mg; ≥50 kg and < 80 kg received 75 mg and ≥ 80 kg and ≤ 150 kg received 150 mg of aliskiren.
  During Phase 2: 30 participants continued the aliskiren treatment from Phase 1, while 21 participants switched to placebo treatment.
- Aliskiren High (150/300/600 mg): During Phase 1: Participants received body-weight stratified dose of aliskiren capsules (150/300/600 mg) once daily. Participants whose body weight ≥ 20 kg to < 50 kg received 150 mg; ≥50 kg and < 80 kg received 300 mg and ≥ 80 kg and ≤ 150 kg received 600 mg of aliskiren.
  During Phase 2: 50 participants continued the aliskiren treatment from Phase 1, while 52 participants switched to placebo treatment.
Period: Dose Response Phase (Phase 1)
Arm/Group | Aliskiren Low (6.25/12.5/25 mg) | Aliskiren Mid (37.5/75/150 mg) | Aliskiren High (150/300/600 mg)
Started | 108 | 54 | 105
Completed | 107 | 51 | 102
Not Completed | 1 | 3 | 3
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Unsatisfactory therapeutic effect | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Participants | 0 | 2 | 1
Period: Placebo-controlled Withdrawal (Phase 2)
Arm/Group | Aliskiren Low (6.25/12.5/25 mg) | Aliskiren Mid (37.5/75/150 mg) | Aliskiren High (150/300/600 mg)
Started | 107 | 51 | 102
Started Aliskiren Treament | 50 | 30 | 50
Completed Aliskiren Treament | 50 | 30 | 49
Started Placebo Treatment | 57 | 21 | 52
Completed Placebo Treament | 54 | 21 | 51
Completed | 104 | 51 | 100
Not Completed | 3 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis was performed in the full analysis set population consisted of all participants who were randomized into the study.
Groups:
- Phase 1: Aliskiren Low (6.25/12.5/25 mg): Participants received body-weight stratified dose of aliskiren capsules (6.25/12.5/25 mg) once daily. Participants whose body weight greater than or equal to (≥) 20 kilogram (kg) to less than (< ) 50 kg received 6.25 mg; ≥50 kg and < 80 kg received 12.5 mg and ≥ 80 kg and less than or equal to (≤)150 kg received 25 mg of aliskiren.
- Phase 1: Aliskiren Mid (37.5/75/150 mg): Participants received body-weight stratified dose of aliskiren capsules (37.5/75/150 mg) once daily. Participants whose body weight ≥ 20 kg to < 50 kg received 37.5 mg; ≥50 kg and < 80 kg received 75 mg and ≥ 80 kg and ≤ 150 kg received 150 mg of aliskiren.
- Phase 1: Aliskiren High (150/300/600 mg): Participants received body-weight stratified dose of aliskiren capsules (150/300/600 mg) once daily. Participants whose body weight ≥ 20 kg to < 50 kg received 150 mg; ≥50 kg and < 80 kg received 300 mg and ≥ 80 kg and ≤ 150 kg received 600 mg of aliskiren.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Aliskiren Low (6.25/12.5/25 mg) | Phase 1: Aliskiren Mid (37.5/75/150 mg) | Phase 1: Aliskiren High (150/300/600 mg) | Total
Number analyzed (Participants) | 108 | 54 | 105 | 267
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.9 (3.27) | 11.6 (3.29) | 11.8 (3.5) | 11.8 (3.36)
Age, Customized [Number; unit: participants]
  Children 6 - 11 years | 49 | 28 | 51 | 128
  Adolescents 12 - 17 years | 59 | 26 | 54 | 139
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 17 | 39 | 91
  Male | 73 | 37 | 66 | 176

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (msSBP) at Endpoint (Phase 1)
Description: Sitting blood pressure was measured using a calibrated standard sphygmomanometer after the participants remained in sitting position for 5 minutes at clinic during the visit. The repeat sitting measurements were made at 1-2 minute intervals and the mean of three sSBP measurements were used as the average sitting office blood pressure for that visit.
Time Frame: Baseline to endpoint (Week 4 or Last observation carried forward (LOCF))
Population: The primary analysis was performed on the Full Analysis Set (FAS), defined as all participants who received at least one dose of study treatment and had at least one post-baseline assessment for primary efficacy. Here, "Number of participants analyzed" signifies participants evaluable for msSBP at Week 4 or LOCF for each arm, respectively.
Measure: Mean (Standard Error); unit: millimeter(s) of mercury (mmHg)
Groups:
- Phase 1: Aliskiren Low (6.25/12.5/25 mg): Participants received body-weight stratified dose of aliskiren capsules (6.25/12.5/25 mg) once daily. Participants whose body weight ≥ 20 kilogram (kg) to less than < 50 kg received 6.25 mg; ≥50 kg and < 80 kg received 12.5 mg and ≥ 80 kg and ≤ 150 kg received 25 mg of aliskiren.
Arm/Group | Phase 1: Aliskiren Low (6.25/12.5/25 mg) | Phase 1: Aliskiren Mid (37.5/75/150 mg) | Phase 1: Aliskiren High (150/300/600 mg)
Number analyzed (Participants) | 108 | 53 | 104
millimeter(s) of mercury (mmHg) | -5.54 (0.78) | -5.42 (1.331) | -9.03 (1.008)

2. Primary Outcome: Change in Mean Sitting Systolic Blood Pressure (msSBP) From Week 4 to Endpoint (Phase 2)
Description: as for outcome 1
Time Frame: Week 4 to endpoint (Week 8 or LOCF)
Population: The primary analysis was performed on the FAS population.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- Phase 2: Aliskiren Low (6.25/12.5/25 mg): Participants received body-weight stratified dose of aliskiren capsules (6.25/12.5/25 mg) once daily. Participants whose body weight ≥ 20 kg to < 50 kg received 6.25 mg; ≥50 kg and < 80 kg received 12.5 mg and ≥ 80 kg and ≤ 150 kg received 25 mg of aliskiren.
- Phase 2: Placebo Low: Participants received placebo capsules matching to aliskiren capsules (6.25/12.5/25 mg) once daily.
- Phase 2: Aliskiren Mid (37.5/75/150 mg): Participants received body-weight stratified dose of aliskiren capsules (37.5/75/150 mg) once daily. Participants whose body weight ≥ 20 kg to < 50 kg received 37.5 mg; ≥50 kg and < 80 kg received 75 mg and ≥ 80 kg and ≤ 150 kg received 150 mg of aliskiren.
- Phase 2: Placebo Mid: Participants received placebo capsules matching to aliskiren capsules (37.5/75/150 mg) once daily.
- Phase 2: Aliskiren High (150/300/600 mg): Participants received body-weight stratified dose of aliskiren capsules (150/300/600 mg) once daily. Participants whose body weight ≥ 20 kg to < 50 kg received 150 mg; ≥50 kg and < 80 kg received 300 mg and ≥ 80 kg and ≤ 150 kg received 600 mg of aliskiren.
- Phase 2: Placebo High: Participants received placebo capsules matching to aliskiren capsules (150/300/600 mg) once daily.
Arm/Group | Phase 2: Aliskiren Low (6.25/12.5/25 mg) | Phase 2: Placebo Low | Phase 2: Aliskiren Mid (37.5/75/150 mg) | Phase 2: Placebo Mid | Phase 2: Aliskiren High (150/300/600 mg) | Phase 2: Placebo High
Number analyzed (Participants) | 50 | 57 | 30 | 21 | 49 | 52
mmHg | -0.53 (0.947) | -0.64 (1.256) | -2.59 (1.119) | -2.9 (1.481) | -1.97 (1.071) | 1.11 (1.185)

3. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events From Baseline to Week 4 (Phase 1)
Description: Adverse events (AEs) were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events (SAEs) were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards.
Time Frame: Baseline up to Week 4
Population: The analysis was performed on the Safety Sets (SAF), SAF is all participants who received at least one dose of study treatment during phase 1 (baseline to week 4)
Measure: Number; unit: participants
Arm/Group | Phase 1: Aliskiren Low (6.25/12.5/25 mg) | Phase 1: Aliskiren Mid (37.5/75/150 mg) | Phase 1: Aliskiren High (150/300/600 mg)
Number analyzed (Participants) | 108 | 54 | 105
participants
  AEs | 30 | 14 | 37
  SAEs | 0 | 0 | 1

4. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events From Week 4 to Week 8 (Phase 2)
Description: AEs were defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. SAEs were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards.
Time Frame: From Week 4 to Week 8
Population: The analysis was performed on the SAF which included all participants who received at least one dose of study treatment during phase 2 (week 4 to week 8).
Measure: Number; unit: participants
Arm/Group | Phase 2: Aliskiren Low (6.25/12.5/25 mg) | Phase 2: Placebo Low | Phase 2: Aliskiren Mid (37.5/75/150 mg) | Phase 2: Placebo Mid | Phase 2: Aliskiren High (150/300/600 mg) | Phase 2: Placebo High
Number analyzed (Participants) | 50 | 57 | 30 | 21 | 50 | 52
participants
  AEs | 18 | 22 | 10 | 5 | 21 | 17
  SAEs | 0 | 0 | 0 | 0 | 2 | 0

5. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (msDBP) at Endpoint (Phase 1)
Description: Sitting blood pressure was measured using a calibrated standard sphygmomanometer after the participants remained in sitting position for 5 minutes at clinic during the visit. The repeat sitting measurements were made at 1-2 minute intervals and the mean of three sDBP measurements were used as the average sitting office blood pressure for that visit.
Time Frame: Baseline to endpoint (Week 4 or LOCF)
Population: The analysis was performed on the FAS population. Here, "Number of participants analyzed" signifies participants evaluable for msDBP at Week 4 or LOCF for each arm, respectively.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Phase 1: Aliskiren Low (6.25/12.5/25 mg) | Phase 1: Aliskiren Mid (37.5/75/150 mg) | Phase 1: Aliskiren High (150/300/600 mg)
Number analyzed (Participants) | 108 | 53 | 104
mmHg | -2.71 (0.67) | -4.05 (1.116) | -6.33 (0.793)

6. Secondary Outcome: Change in Mean Sitting Diastolic Blood Pressure (msDBP) From Week 4 to Endpoint (Phase 2)
Description: as for outcome 5
Time Frame: Week 4 to endpoint (Week 8 or LOCF)
Population: The analysis was performed on the FAS population. Here, "Number of participants analyzed" signifies participants evaluable for msDBP at Week 8 or LOCF for each arm, respectively.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Phase 2: Aliskiren Low (6.25/12.5/25 mg) | Phase 2: Placebo Low | Phase 2: Aliskiren Mid (37.5/75/150 mg) | Phase 2: Placebo Mid | Phase 2: Aliskiren High (150/300/600 mg) | Phase 2: Placebo High
Number analyzed (Participants) | 50 | 57 | 30 | 21 | 49 | 52
mmHg | 1.27 (1.025) | -1.08 (1.012) | 0.89 (1.502) | 1.52 (1.248) | 0.37 (1.052) | 1.51 (1.009)

7. Secondary Outcome: Change From Baseline in Mean Arterial Pressure (MAP) at Endpoint (Phase 1)
Description: MAP was defined as the average arterial pressure during a single cardiac cycle. The MAP was measured as sum of diastolic blood pressure (DBP) and one third of difference between systolic blood pressure (SBP) and DBP i.e. MAP = DBP+1/3*(SBP-DBP).
Time Frame: Baseline to endpoint (Week 4 or LOCF)
Population: The analysis was performed on the FAS population. Here, "Number of participants analyzed" signifies participants evaluable for MAP at Week 4 (or LOCF) for each arm, respectively.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Phase 1: Aliskiren Low (6.25/12.5/25 mg) | Phase 1: Aliskiren Mid (37.5/75/150 mg) | Phase 1: Aliskiren High (150/300/600 mg)
Number analyzed (Participants) | 108 | 53 | 104
mmHg | -3.65 (0.613) | -4.51 (1.064) | -7.23 (0.711)

8. Secondary Outcome: Change in Mean Arterial Pressure (MAP) From Week 4 to Endpoint (Phase 2)
Description: MAP was defined as the average arterial pressure during a single cardiac cycle. The MAP was measured as sum of DBP and one third of difference between SBP and DBP i.e. MAP = DBP+1/3*(SBP-DBP).
Time Frame: Week 4 to endpoint (Week 8 or LOCF)
Population: The analysis was performed on the FAS population. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Phase 2: Aliskiren Low (6.25/12.5/25 mg) | Phase 2: Placebo Low | Phase 2: Aliskiren Mid (37.5/75/150 mg) | Phase 2: Placebo Mid | Phase 2: Aliskiren High (150/300/600 mg) | Phase 2: Placebo High
Number analyzed (Participants) | 50 | 57 | 30 | 21 | 49 | 52
mmHg | 0.67 (0.864) | -0.93 (0.964) | -0.27 (1.239) | 0.05 (1.14) | -0.41 (0.885) | 1.37 (0.918)

9. Secondary Outcome: Percentage of Participants Achieving a Positive Treatment Response at Endpoint (Phase 1)
Description: Treatment responders were defined as participants with msSBP less than 95th percentile (for age, gender and height) or a 7 mmHg decrease in msSBP from the baseline.
Time Frame: Baseline to endpoint (Week 4 or LOCF)
Population: The analysis was performed on the FAS population. Here, "Number of participants analyzed" signifies participants evaluable for this outcome measure at Week 4 or LOCF for each arm, respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | Phase 1: Aliskiren Low (6.25/12.5/25 mg) | Phase 1: Aliskiren Mid (37.5/75/150 mg) | Phase 1: Aliskiren High (150/300/600 mg)
Number analyzed (Participants) | 108 | 53 | 104
Percentage of participants | 50.9 | 58.5 | 69.2

10. Secondary Outcome: Change From Baseline in Mean Ambulatory Systolic and Diastolic Blood Pressure (MASBP and MADBP) at Endpoint (Phase 1)
Description: Ambulatory Blood Pressure Monitoring (ABPM) was performed over a 24-hour period using an automatic ABPM device to record the blood pressure as per study defined criteria. The participants who were selected for this evaluation wore the ABPM device for 24 hours, returned to the clinic upon completion of the 24-hour monitoring period for removal of device and BP assessments. The ABPM device was pre-set to collect readings every 20 minutes. Mean hourly systolic and diastolic blood pressure were calculated for each participant at post dosing 1 - 24 hours.
Time Frame: Baseline to endpoint (Week 4 or LOCF)
Population: Analysis was performed in subset of FAS participants from selected centers who consented to undergo ABPM at baseline and at Week 4 or LOCF. Here 'Number of participants analyzed' signifies those participants evaluable for this measure at specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phase 1: Aliskiren Low (6.25/12.5/25 mg) | Phase 1: Aliskiren Mid (37.5/75/150 mg) | Phase 1: Aliskiren High (150/300/600 mg)
Number analyzed (Participants) | 58 | 29 | 65
mmHg
  MASBP (n=58, 29, 65) | -1.6 (6.48) | -5.9 (5.8) | -5.8 (7.15)
  MADBP (n=58, 29, 65) | -1.1 (5.33) | -4.4 (4.41) | -4.9 (6.05)

11. Secondary Outcome: Change From Baseline in Mean Ambulatory Systolic Blood Pressure (MASBP) During Day and Night at Week 4 (Phase 1)
Description: ABPM was performed over a 24-hour period using an automatic ABPM device to record the blood pressure as per study defined criteria. Day time was defined as the average of the hourly means between 6 am and 10 pm while the night time mean was the average of the hourly means between 10 pm and 6 am.
Time Frame: Baseline to Week 4
Population: Analysis was performed in subset of FAS participants from selected centers who consented to undergo ABPM at baseline and at Week 4. The 'n' signifies those participants evaluable for this measure at specified time points for each group, respectively.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Phase 1: Aliskiren Low (6.25/12.5/25 mg) | Phase 1: Aliskiren Mid (37.5/75/150 mg) | Phase 1: Aliskiren High (150/300/600 mg)
Number analyzed (Participants) | 58 | 29 | 65
mmHg
  Day time (n= 58, 29, 65) | -2.72 (1.031) | -6.76 (1.381) | -6.56 (0.95)
  Night time (n= 57, 29, 65) | -2.55 (1.035) | -4.67 (1.381) | -4.9 (0.95)

12. Secondary Outcome: Change From Baseline in Mean Ambulatory Blood Pressure (MABP) in Dipper Participants at Endpoint (Phase 1)
Description: ABPM was performed over a 24-hour period using an automatic ABPM device to record the blood pressure as per study defined criteria. Dippers were defined as those participants in whom there was a decrease in mean night time (6pm - 6am) ABPM more than or equal to (≥ ) 10% as compared to average daytime (6am -6pm) ABPM.
Time Frame: Baseline to endpoint (Week 4 or LOCF)
Population: Analysis was performed in subset of FAS participants from selected centers who consented to undergo ABPM at baseline and at Week 4 or LOCF. Here, "Number of participants analyzed" signifies participants evaluable for this outcome measure at Week 4 or LOCF for each arm, respectively.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phase 1: Aliskiren Low (6.25/12.5/25 mg) | Phase 1: Aliskiren Mid (37.5/75/150 mg) | Phase 1: Aliskiren High (150/300/600 mg)
Number analyzed (Participants) | 40 | 21 | 47
mmHg
  MASBP | -1.2 (6.18) | -4.6 (5.47) | -6 (6.19)
  MADBP | -0.6 (5.78) | -3.6 (4.19) | -5.3 (5.55)

13. Secondary Outcome: Change From Baseline in Mean Ambulatory Blood Pressure (MABP) in Non--Dipper Participants at Endpoint (Phase 1)
Description: ABPM was performed over a 24-hour period using an automatic ABPM device to record the blood pressure as per study defined criteria. Non-dippers were defined as those participants in whom there was a decrease in mean night time ABPM less than 10% as compared to average daytime ABPM.
Time Frame: Baseline to endpoint (Week 4 or LOCF)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phase 1: Aliskiren Low (6.25/12.5/25 mg) | Phase 1: Aliskiren Mid (37.5/75/150 mg) | Phase 1: Aliskiren High (150/300/600 mg)
Number analyzed (Participants) | 18 | 8 | 18
mmHg
  MASBP | -2.6 (7.21) | -9.3 (5.54) | -5.2 (9.39)
  MADBP | -2.3 (4.05) | -6.7 (4.45) | -5.2 (7.3)

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Participant First Visit (FPFV) Baseline up to 8 weeks until Last Participant Last Visit (LPLV). All adverse events reported in this record are from date of First Participant First Treatment until LPLV.
Groups:
- Phase 1: Aliskiren Low (6.25/12.5/25 mg); Phase 2: Aliskiren Low (6.25/12.5/25 mg): Participants received bodyweight stratified dose of aliskiren capsules (6.25/12.5/25 mg) once daily. Participants whose body weight ≥ 20 kg to < 50 kg received 6.25 mg; ≥50 kg and < 80 kg received 12.5 mg and ≥ 80 kg and ≤ 150 kg received 25 mg of aliskiren.
- Phase 1: Aliskiren Mid (37.5/75/150 mg); Phase 2: Aliskiren Mid (37.5/75/150 mg): Participants received bodyweight stratified dose of aliskiren capsules (37.5/75/150 mg) once daily. Participants whose body weight ≥ 20 kg to < 50 kg received 37.5 mg; ≥50 kg and < 80 kg received 75 mg and ≥ 80 kg and ≤ 150 kg received 150 mg of aliskiren.
- Phase 1: Aliskiren High (150/300/600 mg); Phase 2: Aliskiren High (150/300/600 mg): Participants received bodyweight stratified dose of aliskiren capsules (150/300/600 mg) once daily. Participants whose body weight ≥ 20 kg to < 50 kg received 150 mg; ≥50 kg and < 80 kg received 300 mg and ≥ 80 kg and ≤ 150 kg received 600 mg of aliskiren.
- Phase 2: Placebo Mid: Participants received placebo capsules matching to aliskiren capsules(37.5/75/150 mg) once daily.
Arm/Group | Phase 1: Aliskiren Low (6.25/12.5/25 mg) | Phase 1: Aliskiren Mid (37.5/75/150 mg) | Phase 1: Aliskiren High (150/300/600 mg) | Phase 2: Aliskiren Low (6.25/12.5/25 mg) | Phase 2: Aliskiren Mid (37.5/75/150 mg) | Phase 2: Aliskiren High (150/300/600 mg) | Phase 2: Placebo Low | Phase 2: Placebo Mid | Phase 2: Placebo High
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/54 | 1/105 | 0/50 | 0/30 | 2/50 | 0/57 | 0/21 | 0/52
Other Adverse Events (participants affected / at risk) | 11/108 | 6/54 | 14/105 | 8/50 | 7/30 | 9/50 | 7/57 | 3/21 | 5/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Aliskiren Low (6.25/12.5/25 mg) (N=108) | Phase 1: Aliskiren Mid (37.5/75/150 mg) (N=54) | Phase 1: Aliskiren High (150/300/600 mg) (N=105) | Phase 2: Aliskiren Low (6.25/12.5/25 mg) (N=50) | Phase 2: Aliskiren Mid (37.5/75/150 mg) (N=30) | Phase 2: Aliskiren High (150/300/600 mg) (N=50) | Phase 2: Placebo Low (N=57) | Phase 2: Placebo Mid (N=21) | Phase 2: Placebo High (N=52)
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Aliskiren Low (6.25/12.5/25 mg) (N=108) | Phase 1: Aliskiren Mid (37.5/75/150 mg) (N=54) | Phase 1: Aliskiren High (150/300/600 mg) (N=105) | Phase 2: Aliskiren Low (6.25/12.5/25 mg) (N=50) | Phase 2: Aliskiren Mid (37.5/75/150 mg) (N=30) | Phase 2: Aliskiren High (150/300/600 mg) (N=50) | Phase 2: Placebo Low (N=57) | Phase 2: Placebo Mid (N=21) | Phase 2: Placebo High (N=52)
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 5 | 3 | 3 | 4 | 2 | 1 | 2
Headache (Nervous system disorders) | 5 | 3 | 7 | 4 | 1 | 4 | 3 | 2 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 2 | 2 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.